CLINICAL TRIAL: NCT01677182
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Once a Day, TAK-375 (Ramelteon) Tablet for Sublingual Administration (TAK-375SL Tablet) as an Adjunctive Therapy in the Treatment of Acute Depressive Episodes Associated With Bipolar 1 Disorder in Adult Subjects
Brief Title: Safety and Efficacy Study of Ramelteon (TAK-375) Tablets for Sublingual Administration (SL) in Adults With Bipolar 1 Disorder
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business Decision; Terminated due to futility, with no safety concerns (see below)
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-375SL_301; 2012-001357-10 (EudraCT Number); U1111-1129-5184 (Registry Identifier: WHO); 12/EM/0391 (Registry Identifier: NRES)
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Results first posted 2016-03-16 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-02

CONDITIONS: Bipolar Disorder
Keywords: Drug therapy
MeSH Terms: conditions — Bipolar Disorder | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ramelteon SL (Dose 1) (Experimental): Ramelteon SL tablets, sublingual, once daily, at night time for up to 6 weeks.
  Interventions: Drug: Ramelteon
- Ramelteon (Dose 2) (Experimental): Ramelteon SL tablets, sublingual, once daily, at night time for up to 6 weeks.
  Interventions: Drug: Ramelteon
- Placebo (Placebo Comparator): Ramelteon SL placebo-matching tablets, sublingual, once daily, at night time for up to 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon — Ramelteon tablets for sublingual administration
  Other Names: TAK-375SL; Rozerem
  Arms: Ramelteon (Dose 2); Ramelteon SL (Dose 1)
Drug: Placebo — Ramelteon placebo-matching tablets for sublingual administration
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of ramelteon for treatment of acute depressive episodes associated with Bipolar 1 Disorder.

DETAILED DESCRIPTION:
The drug being tested in this study is called Ramelteon. Ramelteon is being tested to treat people who have Bipolar 1 Disorder. This study will look at the symptoms of depression in people who take Ramelteon as a sub-lingual formulation.

This study plans to enroll a minimum of 276 participants and a maximum of up to approximately 870 participants Participants will be randomly assigned (by chance, like flipping a coin) to one of the three treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* Ramelteon (Dose 1)
* Ramelteon (Dose 2)
* Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient All participants will be asked to take one tablet every night at bedtime throughout the study.

This study plans to conduct one unblinded interim analysis after the first 276 subjects have been enrolled and treated for the 6-week double-blind treatment period. Based on the interim analysis, the study plans to adapt limited aspects of the design including: 1) to make no changes to the study; 2) to reassess sample size based on the interim analysis results.

This multi-centre trial will be conducted in North America and Europe. The overall time to participate in this study is up to 14 weeks. Participants will make 8 visits to the clinic, and will be contacted by telephone 30 days after last dose of study drug for a follow-up assessment.

An independent Data Monitoring Committee (DMC) recently performed a planned interim analysis of efficacy and safety data from this study. Upon completion of their review, the DMC advised that the unblinded interim data met the predefined efficacy criteria for study termination. No safety concerns were identified.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the subject is capable of understanding and complying with protocol requirements.
2. The subject or, when applicable, the subject's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. The subject suffers from Bipolar 1 Disorder, Most Recent Episode Depressed as the primary diagnosis according to DSM-IV-TR criteria (classification code 296.5x) and confirmed by the SCID.
4. The subject is a man or woman aged between 18 and 75 years, inclusive.
5. The reported duration of the current Major Depressive Episode (MDE) is at least four weeks and less than 6 months.
6. The subject has a YMRS total score of ≤10 both at the Screening and Baseline Visits.
7. The subject has a MADRS total score of ≥24 at the Screening and Baseline Visits.
8. The subject has a CGI-S score of ≥4 at the Screening and Baseline Visits.
9. The subject has HAM- A total score of ≤21 at Screening and Baseline Visits.
10. The subject is on lithium and/or one other mood stabilizer (lamotrigine or valproic acid) and/or one atypical antipsychotic (risperidone or olanzapine or aripiprazole or ziprasidone). Patients may be on one, two, or three medications but no more than one from each group.
11. The subject is on the same dose of the protocol allowed medications (identified in inclusion # 10) for bipolar 1 disorder for at least two weeks prior to screening (and at least 6 weeks prior to screening for lamotrigine only). Further dose adjustments will not be allowed from screening until end of study, except for downward dose adjustments for adverse events.
12. If the subject is on lithium and/or valproic acid, the trough serum levels must be less than 1.2 mEq/L for lithium and the trough serum must be less than 125 mcg/ml for valproic acid. Downward dose adjustment is allowed to lower trough serum levels for lithium and/or valproic acid below the maximum allowed. This must be confirmed at least two weeks prior to baseline.
13. The subject screened must have <25% improvement in MADRS total score from screening to baseline visit with a minimum of two weeks between screening and baseline visits.
14. A female subject of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study and for 30 days after the last dose of the study drug.
15. A male subject who is nonsterilized and sexually active with female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 30 days after the last dose of study drug.

Exclusion Criteria:

1. The subject has received any investigational compound <30 days before Screening or 5 half-lives whichever is longer prior to Screening.
2. The subject has received TAK-375 or TAK-375SL in a previous clinical study or has ever used ramelteon.
3. The subject is an immediate family member, study site employee, or is in a dependant relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
4. The subject has one or more of the following:

   1. Any current psychiatric disorder which is the primary focus of treatment other than Bipolar 1 Disorder, Most Recent Episode Depressed as defined in the DSM-IV-TR, as assessed by the SCID.
   2. Current or history of: schizophrenia, schizoaffective disorder, unipolar depression with psychotic features, bipolar depression with psychotic features, any other psychotic disorder (with the exception of psychosis associated with a manic or mixed episode), mental retardation, organic mental disorders, OCD, or mental disorders due to a general medical condition as defined in the DSM-IV-TR.
   3. Current diagnosis or history of alcohol or other substance abuse (excluding nicotine or caffeine) as defined in the DSM-IV-TR that has not been in full and sustained remission for at least three months from the day of screening. (Subject must also have negative urine drug screen at Screening and Baseline). Note that a positive drug screen for opiates and benzodiazepines is allowed provided the subject has a valid prescription.
   4. Current diagnosis or history of alcohol or other substance dependence (excluding nicotine or caffeine) as defined in the DSM-IV-TR that has not been in full and sustained remission for at least three months from the day of screening. (Subject must also have negative urine drug screen at screening and Baseline). Note that a positive drug screen for opiates and benzodiazepines is allowed provided the subject has a valid prescription.
   5. Presence or history of a clinically significant neurological disorder (including epilepsy).
   6. Neurodegenerative disorder (Alzheimer disease, Parkinson disease, multiple sclerosis, Huntington disease, etc).
   7. Any Axis II disorder that might compromise the study.
   8. History of Rapid Cycling Bipolar Disorder: Patients who have more than 8 episodes of mood disorder per year. The episodes must meet both the duration and symptom criteria for a major depressive, manic, mixed, or hypomanic episode and must be demarcated by either a period of full remission or by a switch to an episode of the opposite polarity. manic, hypomanic, and mixed episodes are counted as being on the same pole. Each mood episode must be confirmed by appropriate patient history or formal diagnosis by medical practitioner.
5. The subject experienced the first episode of mood disorder after the age of 55 years.
6. The current depressive symptoms of the subject are considered by the investigator to have been resistant to 2 adequate treatment trials with any of the mood stabilizers (specifically started to treat the current depressive episode) and/or medications approved for acute bipolar depression (e.g. quetiapine, olanzapine + fluoxetine [US only]) for at least 6 weeks duration each.
7. The subject is on any psychotropic medications other than the protocol allowed medications for at least 2 weeks prior to the Baseline visit. If a subject is taking any protocol excluded medications (e.g. antidepressants, typical antipsychotics) or is taking more than one of the allowed mood stabilizer and/or atypical antipsychotic medications, and if the patient is considered appropriate by the PI, these medications must be washed out for at least 2 weeks prior to the Baseline visit.
8. The subject has received electroconvulsive therapy, vagal nerve stimulation, or repetitive transcranial magnetic stimulation within 6 months prior to Screening.
9. The subject has started receiving formal cognitive or behavioral therapy, systematic psychotherapy within 30 days prior to screening or plans to initiate such therapy during the study.
10. The subject has a significant risk of suicide according to the investigator's clinical judgment or has a score ≥5 on item 10 (suicidal thoughts) of the MADRS or has made a suicide attempt in the previous 6 months.
11. The subject has taken or is anticipated that the subject will take at least 1 of the disallowed concomitant medications that is listed in the Excluded Medications and Treatments (Table 7.a).
12. The subject has a clinically significant unstable illness, for example hepatic impairment or renal insufficiency, or a cardiovascular, pulmonary, gastrointestinal, endocrine, neurological, rheumatologic, immunologic, hematological, infectious, dermatological disorder or metabolic disturbance as determined by Investigator.
13. The subject has a history or current diagnosis of fibromyalgia, chronic fatigue syndrome, chronic pain syndrome or sleep apnea (central and/or obstructive). If obstructive sleep apnea is corrected surgically, a polysomnogram showing normal apnea-hypopnea index is required.
14. The subject has a previous history of cancer that had been in remission for less than 5 years prior to the first dose of study medication. This criterion does not include those subjects with basal cell or stage I squamous cell carcinoma of the skin.
15. The subject has 1 or more laboratory value outside the normal range, based on the blood or urine samples taken at the Screening Visit, that are considered by the investigator to be clinically significant; or the subject has any of the following values at the Screening Visit:

    1. A serum creatinine value >1.5 times the upper limits of normal (xULN).
    2. A serum total bilirubin value >1.5 xULN.
    3. A serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value >2 xULN.
16. The subject has HbA1C ≥7% at screening and no prior diagnosis of diabetes and/or treatment for diabetes. NOTE: Subjects with known diabetes are not excluded.
17. The subject has a thyroid stimulating hormone (TSH) value outside the normal range at the Screening Visit that is deemed clinically significant by the investigator. NOTE: Free thyroxine (T4) will be checked if TSH is out of range. If free T4 is abnormal the subject will be excluded.
18. The subject is positive for hepatitis B surface antigen (HBsAg), antibodies to hepatitis C virus (HCV), or has a history of human immunodeficiency virus (HIV) infection.
19. If male, the subject intends to donate sperm during the course of this study or for 12 weeks thereafter. If female, the subject is pregnant or lactating or intending to become pregnant before, during, or within 30 days after participating in this study; or intending to donate ova during such time period.
20. The subject has clinically significant abnormal vital signs as determined by the investigator.
21. The subject has an abnormal ECG as determined by the central reader and confirmed as clinically significant by the investigator.
22. The subject has a disease or takes medication that, in the opinion of the investigator, could interfere with the assessments of safety, tolerability, or efficacy.
23. The subject, in the opinion of the investigator, is unlikely to comply with the clinical study protocol or is unsuitable for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda Global Research and Development Center, Inc.
Locations (104):
- United States (41):
  - Birmingham, Alabama
  - Anaheim, California
  - Glendale, California
  - Imperial, California
  - Los Angeles, California
  - Oakland, California
  - Oceanside, California
  - Pico Rivera, California
  - San Diego, California
  - Stanford, California
  - Hartford, Connecticut
  - Coral Springs, Florida
  - Deerfield Beach, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Maitland, Florida
  - Oakland Park, Florida
  - Orlando, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Chicago, Illinois
  - Joliet, Illinois
  - Naperville, Illinois
  - Oak Brook, Illinois
  - Lafayette, Indiana
  - Boston, Massachusetts
  - St Louis, Missouri
  - Buffalo, New York
  - New York, New York
  - Staten Island, New York
  - The Bronx, New York
  - Avon Lake, Ohio
  - Cincinnati, Ohio
  - Garfield Heights, Ohio
  - Mason, Ohio
  - Oklahoma City, Oklahoma
  - Memphis, Tennessee
  - San Antonio, Texas
  - Bothell, Washington
  - Spokane, Washington
  - Waukesha, Wisconsin
- Bulgaria (10):
  - Burgas
  - Kazanlak
  - Lovech
  - Novi Iskar
  - Pleven
  - Plovdiv
  - Rousse
  - Sofia
  - Tzerova Koria
  - Varna
- Czechia (5):
  - Brno
  - Litoměřice
  - Olomouc
  - Pilsen
  - Prague
- Germany (4):
  - Bochum, North Rhine-Westphalia
  - Berlin, State of Berlin
  - Berlin
  - Westerstede
- Poland (2):
  - Bialystok
  - Choroszcz
- Romania (11):
  - Oradea, Bihor County
  - Cluj-Napoca, Cluj
  - Craiova, Dolj
  - Târgovişte, Dâmbovița County
  - Bucharest, Romania
  - Arad
  - Bucharest
  - Cluj-Napoca
  - Craiova
  - Iași
  - Târgovişte
- Russia (11):
  - Talagi, Arkhangelskaya oblast
  - Orenburg, Orenburg Oblast
  - Staritsa Settlement, Orenburg Oblast
  - Saint Petersburg, Sankt-Peterburg
  - Town. Tonnelniy, Stavropol Region
  - Arkhangelsk
  - Moscow
  - Nizhny Novgorod
  - Saint Petersburg
  - Smolensk
  - Stavropol
- Serbia (7):
  - Belgrade, Serbia
  - Kragujevac, Sumadija
  - Novi Sad, Vojvodina
  - Belgrade
  - Kragujevac
  - Niš
  - Novi Kneževac
- Ukraine (9):
  - Simferopol, Autonomous Republic of Crimea
  - Oleksandrivka, Kominternivske District, Odesa Oblast
  - Simferopol, The Autonomous Republic of Crimea
  - Vinnytsia, Vinnytsia Oblast
  - Kharkiv
  - Luhansk
  - Odesa
  - Poltava
  - Ternopil
- United Kingdom (4):
  - Oxford, Oxfordshire
  - Birmingham
  - London
  - Newcastle upon Tyne

REFERENCES:
- See also: Rozerem Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ROZEREMPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part at 98 sites in Bulgaria, the Czech Republic, Germany, Great Britain, Poland, Romania, Russia, Serbia, Ukraine, and the United States from 29 August 2012 to 03 September 2014.
Pre-assignment Details: Participants with a historical diagnosis of bipolar 1 disorder were enrolled in 1 of 3 treatment groups as follows: placebo; TAK-375 0.1 milligram (mg); TAK-375 0.4 mg.
Groups:
- Placebo: TAK-375SL (ramelteon) placebo-matching tablet, sublingually, once daily for up to 6 weeks.
- TAK-375SL 0.1 mg: TAK-375SL (ramelteon) 0.1 mg, tablet, sublingually, once daily for up to 6 weeks.
- TAK-375SL 0.4 mg: TAK-375SL (ramelteon) 0.4 mg, tablet, sublingually, once daily for up to 6 weeks.
Period: Overall Study
Arm/Group | Placebo | TAK-375SL 0.1 mg | TAK-375SL 0.4 mg
Started | 184 | 169 | 182
Completed | 150 | 141 | 143
Not Completed | 34 | 28 | 39
Not completed — Adverse Event | 2 | 1 | 8
Not completed — Protocol Violation | 5 | 1 | 4
Not completed — Lost to Follow-up | 4 | 0 | 3
Not completed — Withdrawal by Subject | 7 | 12 | 10
Not completed — Study termination | 12 | 9 | 11
Not completed — Lack of Efficacy | 3 | 0 | 1
Not completed — Other reasons | 1 | 5 | 2

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | TAK-375SL 0.1 mg | TAK-375SL 0.4 mg | Total
Number analyzed (Participants) | 184 | 169 | 182 | 535
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.67 (11.332) | 45.44 (11.490) | 44.87 (11.608) | 45.67 (11.480)
Age, Customized [Number; unit: participants]
  Less than or equal to (<=) 50 years | 105 | 100 | 107 | 312
  Greater than (>) 50 years | 79 | 69 | 75 | 223
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 98 | 108 | 325
  Male | 65 | 71 | 74 | 210
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 10 | 9 | 31
  Not Hispanic or Latino | 63 | 61 | 63 | 187
  Unknown or Not Reported | 109 | 98 | 110 | 317
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 1 | 3
  Black or African American | 11 | 12 | 12 | 35
  White | 171 | 154 | 166 | 491
  More than one race | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Bulgaria | 31 | 27 | 30 | 88
  Czech Republic | 9 | 7 | 8 | 24
  Germany | 3 | 5 | 3 | 11
  United Kingdom | 1 | 0 | 0 | 1
  Poland | 2 | 4 | 4 | 10
  Romania | 8 | 7 | 9 | 24
  Russian Federation | 12 | 9 | 13 | 34
  Serbia | 22 | 20 | 25 | 67
  Ukraine | 20 | 19 | 18 | 57
  United States | 76 | 71 | 72 | 219
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 168.86 (9.227) | 170.66 (8.423) | 169.80 (8.870) | 169.75 (8.871)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 80.82 (23.503) | 83.21 (18.638) | 82.38 (19.202) | 82.11 (20.605)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 28.25 (7.583) | 28.57 (6.130) | 28.52 (6.156) | 28.44 (6.663)
Smoking Classification [Number; unit: participants]
  Had Never Smoked | 84 | 75 | 79 | 238
  Current Smoker | 75 | 70 | 82 | 227
  Ex-smoker | 25 | 24 | 21 | 70
Subject Drinking Status [Number; unit: participants]
  Had Never Drunk | 97 | 92 | 109 | 298
  Ex-Drinker | 51 | 41 | 36 | 128
  Current Drinker | 36 | 36 | 37 | 109
Amount of Alcohol Consumed if Current Drinker [Number; unit: participants] — Participants evaluable for this measure included only those who were current drinkers (36, 36, and 37 for each group, respectively).
  participants
    < 4 drinks per day | 36 | 36 | 37 | 109
    >= 4 drinks per day | 0 | 0 | 0 | 0
Consumption of Caffeine [Number; unit: participants]
  Consumer | 140 | 128 | 144 | 412
  Not a consumer | 44 | 41 | 38 | 123
Psychiatric History for response to Lithium treatment for Bipolar 1 Disorder [Number; unit: participants]
  Failed to Respond | 7 | 7 | 7 | 21
  Responded | 101 | 92 | 100 | 293
  Not Applicable | 69 | 63 | 68 | 200
  Unknown | 7 | 7 | 7 | 21
Psychiatric History for response to Valproic Acid Treatment of Bipolar 1 Disorder [Number; unit: participants]
  Failed to Respond | 6 | 8 | 9 | 23
  Responded | 133 | 124 | 136 | 393
  Not Applicable | 35 | 29 | 27 | 91
  Unknown | 10 | 8 | 10 | 28
Female Reproductive Status [Number; unit: participants]
  Postmenopausal | 44 | 30 | 34 | 108
  Surgically Sterile | 20 | 14 | 12 | 46
  Child-Bearing Potential | 55 | 54 | 62 | 171
  Not applicable (male participants) | 65 | 71 | 74 | 210

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score at Week 6
Description: The MADRS is a clinician rated, validated and widely used scale to measure overall severity of depressive symptoms. It consists of 10-item rated from 0(normal) to 6(most abnormal) with a total score range from 0 to 60. Higher scores indicate greater severity of symptoms.
Time Frame: Baseline and Week 6
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of double-blind study medication and who had a baseline value and at least 1 valid post-baseline value for assessment of primary efficacy.
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | TAK-375SL 0.1 mg | TAK-375SL 0.4 mg
Number analyzed (Participants) | 179 | 167 | 176
units on scale
  Baseline (n= 179, 167, 176) | 30.8 (0.28) | 30.2 (0.29) | 30.4 (0.29)
  Change at Week 6 (n= 149, 139, 143) | -14.7 (0.69) | -14.0 (0.71) | -15.1 (0.70)
Statistical Analysis 1: Comparison: Placebo vs TAK-375SL 0.1 mg; Test type: Superiority or Other; p = 0.783, Mixed Model Repeated Measures — Mixed Model Repeated Measures (MMRM) model with baseline by week interaction, pooled center, week, treatment, baseline, and week by treatment interaction as factors was used for the analysis; Least Squares Mean Differences = 0.8, 97.5% CI 2-sided [-1.4 to 3.0], Standard Error of Mean 0.98
Statistical Analysis 2: Comparison: Placebo vs TAK-375SL 0.4 mg; Test type: Superiority or Other; p = 0.329, Mixed Model Repeated Measures — MMRM model with baseline by week interaction, pooled center, week, treatment, baseline, and week by treatment interaction as factors was used for the analysis; Least Squares Mean Difference = -0.4, 97.5% CI 2-sided [-2.6 to 1.7], Standard Error of Mean 0.97

2. Secondary Outcome: Change From Baseline in Young Mania Rating Scale (YMRS) Total Score at Week 6
Description: The YMRS is a 11-item scale to assess manic symptoms. Four items are rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe), and 7 items are rated on a scale from 0 to 4 with higher scores reflecting greater levels of mania. The YMRS total score is calculated as the sum of the 11 individual item scores and ranges from 0-60.
Time Frame: Baseline and Week 6
Population: FAS included all randomized participants who received at least 1 dose of double-blind study medication and who had a baseline value and at least 1 valid post-baseline value for assessment of primary efficacy.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TAK-375SL 0.1 mg | TAK-375SL 0.4 mg
Number analyzed (Participants) | 179 | 167 | 176
units on a scale
  Baseline (n= 179, 167, 176) | 4.4 (0.16) | 4.3 (0.16) | 4.4 (0.16)
  Change at Week 6 (n= 149, 139, 143) | -1.4 (0.19) | -0.9 (0.20) | -1.5 (0.20)
Statistical Analysis 1: Comparison: Placebo vs TAK-375SL 0.1 mg; Test type: Superiority or Other; p = 0.088, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = 0.5, 97.5% CI 2-sided [-0.1 to 1.1], Standard Error of Mean 0.27
Statistical Analysis 2: Comparison: Placebo vs TAK-375SL 0.4 mg; Test type: Superiority or Other; p = 0.642, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = -0.1, 97.5% CI 2-sided [-0.7 to 0.5], Standard Error of Mean 0.27

3. Secondary Outcome: Clinical Global Impression Scale-Improvement (CGI-I) Score
Description: The CGI-I assesses the clinician's impression of the participant's state of mental illness improvement and consists of 1 question for the investigator: "Compared to his condition at the start of the study, how much has this patient changed?" which is rated on a 7-point scale (1=very much improved; 2=much improved; 3=minimally improved; 4=no change relative to baseline; 5=minimally worse; 6= much worse; 7=very much worse). In all cases, the assessment was independent of whether the rater believed the improvement was drug-related or not.
Time Frame: Week 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TAK-375SL 0.1 mg | TAK-375SL 0.4 mg
Number analyzed (Participants) | 149 | 139 | 143
units on a scale | 2.5 (0.08) | 2.5 (0.09) | 2.3 (0.09)
Statistical Analysis 1: Comparison: Placebo vs TAK-375SL 0.1 mg; Test type: Superiority or Other; p = 0.792, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = 0.0, 97.5% CI 2-sided [-0.2 to 0.3], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Placebo vs TAK-375SL 0.4 mg; Test type: Superiority or Other; p = 0.171, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = -0.2, 97.5% CI 2-sided [-0.4 to 0.1], Standard Error of Mean 0.12

4. Secondary Outcome: Change From Baseline in Clinical Global Impression Scale-Severity (CGI-S) to Week 6
Description: The CGI-S assesses the clinician's impression of the participant's current state of mental illness and consists of 1 question for the investigator: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" which is rated on a 7-point scale (1=normal, not ill at all; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill).
Time Frame: Baseline and Week 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TAK-375SL 0.1 mg | TAK-375SL 0.4 mg
Number analyzed (Participants) | 179 | 167 | 176
units on a scale
  Baseline (n= 179, 167, 176) | 4.5 (0.04) | 4.5 (0.04) | 4.5 (0.04)
  Change at Week 6 (n= 149, 139, 143) | -1.4 (0.08) | -1.3 (0.09) | -1.4 (0.08)
Statistical Analysis 1: Comparison: Placebo vs TAK-375SL 0.1 mg; Test type: Superiority or Other; p = 0.653, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = 0.1, 97.5% CI 2-sided [-0.2 to 0.3], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Placebo vs TAK-375SL 0.4 mg; Test type: Superiority or Other; p = 0.673, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = -0.0, 97.5% CI 2-sided [-0.3 to 0.2], Standard Error of Mean 0.12

5. Secondary Outcome: Change From Baseline in the Quick Inventory of Depressive Symptomatology - Self-Rated16 (QIDS-SR16) Total Score at Week 6
Description: The 16-item QIDS-SR16 version is a widely used validated scale designed to assess the severity of depressive symptoms. The participant was asked to rate the severity and frequency of specific symptoms present over the last 7 days. The QIDS-SR16 total scores range from 0 to 27, where higher scores indicate higher severity of symptoms.
Time Frame: Baseline and Week 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TAK-375SL 0.1 mg | TAK-375SL 0.4 mg
Number analyzed (Participants) | 179 | 167 | 176
units on a scale
  Baseline (n= 178, 167, 176) | 14.8 (0.26) | 14.5 (0.27) | 14.2 (0.26)
  Change at Week 6 (n= 148, 139, 143) | -7.2 (0.36) | -6.4 (0.38) | -7.3 (0.37)
Statistical Analysis 1: Comparison: Placebo vs TAK-375SL 0.1 mg; Test type: Superiority or Other; p = 0.119, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = 0.8, 97.5% CI 2-sided [-0.4 to 2.0], Standard Error of Mean 0.51
Statistical Analysis 2: Comparison: Placebo vs TAK-375SL 0.4 mg; Test type: Superiority or Other; p = 0.791, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = -0.1, 97.5% CI 2-sided [-1.3 to 1.0], Standard Error of Mean 0.51

6. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score at Week 6
Description: The SDS is a 3-item rating scale to assess functional impairment (panic, anxiety, phobic and depressive symptoms) over 3 inter-related domains (work/school, social life, and family life/home responsibilities) rated on an 11-point scale from 0 (not at all) to 10 (extremely) with a total score range from 0 to 30 where higher scores indicates greater severity of impairment.
Time Frame: Baseline and Week 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TAK-375SL 0.1 mg | TAK-375SL 0.4 mg
Number analyzed (Participants) | 179 | 167 | 176
units on a scale
  Baseline (n= 174, 163, 172) | 18.1 (0.43) | 17.1 (0.44) | 15.9 (0.43)
  Change at Week 6 (n= 148, 139, 143) | -6.8 (0.51) | -6.2 (0.52) | -6.4 (0.51)
Statistical Analysis 1: Comparison: Placebo vs TAK-375SL 0.1 mg; Test type: Superiority or Other; p = 0.422, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = 0.6, 97.5% CI 2-sided [-1.0 to 2.1], Standard Error of Mean 0.70
Statistical Analysis 2: Comparison: Placebo vs TAK-375SL 0.4 mg; Test type: Superiority or Other; p = 0.655, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = 0.3, 97.5% CI 2-sided [-1.3 to 1.9], Standard Error of Mean 0.70

7. Secondary Outcome: Change From Baseline in Quality of Life, Enjoyment, and Satisfaction Questionnaire Short Form (Q-LES-Q-SF) Total Score at Week 6
Description: Q-LES-Q-SF is a self-administered, widely used 16-item questionnaire to assess the degree of enjoyment and satisfaction experienced by participants in various areas of daily functioning, such as social relationships, living/housing, physical health, medication, and global satisfaction. The questionnaire consists of 16 items rated by the participants on a 5-point scale. Of these, 14 items are summed to produce a total quality of life score with a maximum of 70 points. In addition, there are 2 global items that are scored individually. These items rate satisfaction with study medication and overall life satisfaction. The questionnaire is usually scored as a percent of the total possible score, with higher scores indicating better health status.
Time Frame: Baseline and Week 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of total possible score
Arm/Group | Placebo | TAK-375SL 0.1 mg | TAK-375SL 0.4 mg
Number analyzed (Participants) | 179 | 167 | 176
percentage of total possible score
  Baseline (n= 174, 163, 172) | 38.3 (0.93) | 38.8 (0.95) | 41.0 (0.93)
  Change at Week 6 (n= 148, 139, 143) | 15.6 (1.19) | 14.7 (1.22) | 15.7 (1.21)
Statistical Analysis 1: Comparison: Placebo vs TAK-375SL 0.1 mg; Test type: Superiority or Other; p = 0.696, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = -0.8, 97.5% CI 2-sided [-4.5 to 2.8], Standard Error of Mean 1.64
Statistical Analysis 2: Comparison: Placebo vs TAK-375SL 0.4 mg; Test type: Superiority or Other; p = 0.472, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = 0.1, 97.5% CI 2-sided [-3.6 to 3.8], Standard Error of Mean 1.63

8. Secondary Outcome: Percentage of Participants With MADRS Response
Description: MADRS response is defined as greater than or equal to (>=) 50 percent (%) decrease in the MADRS total score from baseline. The MADRS is a clinician rated, validated and widely used scale to measure overall severity of depressive symptoms. It consists of 10-item rated from 0 (normal) to 6 (most abnormal) with a total score range from 0 to 60, where higher scores indicate greater severity of symptoms.
Time Frame: Week 6
Population: FAS included all randomized participants who received at least 1 dose of double-blind study medication and who had a baseline value and at least 1 valid post-baseline value for assessment of primary efficacy. Last observation carried forward (LOCF) method was used to impute missing data.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-375SL 0.1 mg | TAK-375SL 0.4 mg
Number analyzed (Participants) | 179 | 167 | 176
percentage of participants | 43.6 | 43.1 | 40.3
Statistical Analysis 1: Comparison: Placebo vs TAK-375SL 0.1 mg; Test type: Superiority or Other; p = 0.994, Regression, Logistic — Odds ratio, 95% confidence intervals and p-values are analyzed from logistic regression with explanatory variables for treatment and baseline MADRS total score; Odds Ratio (OR) = 0.998, 95% CI 2-sided [0.651 to 1.530]
Statistical Analysis 2: Comparison: Placebo vs TAK-375SL 0.4 mg; Test type: Superiority or Other; p = 0.575, Regression, Logistic — [p-value comment as in outcome 8, analysis 1]; Odds Ratio (OR) = 0.886, 95% CI 2-sided [0.580 to 1.352]

9. Secondary Outcome: Percentage of Participants With MADRS Remission
Description: MADRS remission is defined as a MADRS total score less than or equal to (<=) 10. The MADRS is a clinician rated, validated and widely used scale to measure overall severity of depressive symptoms. It consists of 10-item rated from 0 (normal) to 6 (most abnormal) with a total score range from 0 to 60, where higher scores indicate greater severity of symptoms.
Time Frame: Week 6
Population: FAS included all randomized participants who received at least 1 dose of double-blind study medication and who had a baseline value and at least 1 valid post-baseline value for assessment of primary efficacy. LOCF method was used to impute missing data.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-375SL 0.1 mg | TAK-375SL 0.4 mg
Number analyzed (Participants) | 179 | 167 | 176
percentage of participants | 26.8 | 26.9 | 24.4
Statistical Analysis 1: Comparison: Placebo vs TAK-375SL 0.1 mg; Test type: Superiority or Other; p = 0.927, Regression, Logistic — [p-value comment as in outcome 8, analysis 1]; Odds Ratio (OR) = 0.978, 95% CI 2-sided [0.606 to 1.577]
Statistical Analysis 2: Comparison: Placebo vs TAK-375SL 0.4 mg; Test type: Superiority or Other; p = 0.553, Regression, Logistic — [p-value comment as in outcome 8, analysis 1]; Odds Ratio (OR) = 0.865, 95% CI 2-sided [0.536 to 1.397]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 30 days for a serious adverse event after the last dose of double-blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | TAK-375SL 0.1 mg | TAK-375SL 0.4 mg
Serious Adverse Events (participants affected / at risk) | 1/184 | 0/169 | 5/182
Other Adverse Events (participants affected / at risk) | 18/184 | 14/169 | 10/182
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=184) | TAK-375SL 0.1 mg (N=169) | TAK-375SL 0.4 mg (N=182)
Cellulitis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Hypomania (Psychiatric disorders) | 0 | 0 | 1
Mania (Psychiatric disorders) | 0 | 0 | 1
Psychiatric symptom (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=184) | TAK-375SL 0.1 mg (N=169) | TAK-375SL 0.4 mg (N=182)
Headache (Nervous system disorders) | 18 | 14 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.